CLINICAL TRIAL: NCT06734494
Title: Laparoscopic Appendectomy Using Airseal or a Standard Insufflator for Peritonitis in Children
Brief Title: Retrospective Comparison Between AirSeal® and Standard Insufflation in Appendicular Peritonitis
Acronym: APPAS
Status: Completed | Type: Observational
Sponsor: Destinval Christelle (Other)
Responsible Party: Sponsor-Investigator, Destinval Christelle, Dr., University Hospital, Clermont-Ferrand
Organization: University Hospital, Clermont-Ferrand (Other)
Other Study IDs: M24DC1108; NCT05840419 (obsolete NCT alias)
Record Dates: First submitted 2024-12-10; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Peritonitis; Acute; Acute Appendicitis; Postoperative Pain; Laparoscopy
Keywords: Valveless Trocar; Low-pressure Insufflation; Standard insufflation; Laparoscopic Appendectomy; Appendicular Peritonitis; Retrospective Study
MeSH Terms: conditions — Peritonitis; Appendicitis; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Airseal group (A): Patients who underwent a laparoscopic appendectomy using Airseal
  Interventions: Device: Laparoscopic appendectomy Laparoscopic appendectomy with Airseal or with standard insufflation
- Standard group (S): Patients who underwent a laparoscopic appendectomy using standard insufflation
  Interventions: Device: Laparoscopic appendectomy Laparoscopic appendectomy with Airseal or with standard insufflation

INTERVENTIONS:
Device: Laparoscopic appendectomy Laparoscopic appendectomy with Airseal or with standard insufflation — Airseal is a constant and low-pressure insufflation device. Standard insufflation is a variable pressure insufflation device.

SUMMARY:
The AirSeal System Valve-less Trocar is known to decrease postoperative pain, consumption of analgesics, operating time, and length of stay in adults during robotic and laparoscopic procedures. The investigators would like to know if these allegations also apply to children.

DETAILED DESCRIPTION:
From January the 1st 2022 to December the 31st 2022, 100 children aged under 18 years old had an appendicular peritonitis treated by laparoscopic appendectomy. The pediatric surgeons either used the AirSeal System Valve-less Trocar or the standard insufflation. On one hand, only the surgeon, the anesthetist and the nurses of the operating room knew which type of insufflation was used. On the other hand, the patient, his parents and the nurses in the pediatric department did not know which type of insufflation was used. The participants were divided in two groups: the Airseal group (A) and the standard group (S). In each group, the investigators studied and compared the postoperative pain, the consumption of analgesics, the operating time, and the length of stay for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 4 and 17 years old
* Who underwent laparoscopic appendectomy for appendicular peritonitis
* Between 2022/06/1st and 2022/12/31st

Exclusion Criteria:

* Children younger than 4 years old or older than 18 years old
* Who did not have appendicular peritonitis
* Between 2022/01/1st and 2022/12/31st

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients aged between 4 and 17 years old who underwent laparoscopic appendectomy for appendicular peritonitis using the Airseal® or a Standard Insufflation, from 2022/01/1st to 2022/12/31st.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Consumption of analgesics | From the end of surgery to the discharge home, up to 20 days
  Number of medications taken during hospitalization

SECONDARY OUTCOMES:
Length of stay | From the admission to the discharge home, up to 20 days
  Length of stay
Operating Time | From beginning to end of surgery
  Time to operate the patients
Mean Digital Pain Scale | Immediately after surgery until discharge home, up to 20 days
  Digital Pain Scale: minimum is 0 out of 10 (which means no pain) and maximum is 10 out of 10 (which means very painful). Higher scores mean worse outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Clermont-Ferrand, Clermont-Ferrand, Auvergne, France

IPD SHARING:
Plan to Share IPD: No
In the name of anonymization we won't share individual participant data

REFERENCES:
- [Background] Hua J, Gong J, Yao L, Zhou B, Song Z. Low-pressure versus standard-pressure pneumoperitoneum for laparoscopic cholecystectomy: a systematic review and meta-analysis. Am J Surg. 2014 Jul;208(1):143-50. doi: 10.1016/j.amjsurg.2013.09.027. Epub 2014 Jan 16. PMID 24503370
- [Background] Rebuck DA, Zhao LC, Helfand BT, Casey JT, Navai N, Perry KT, Nadler RB. Simple modifications in operating room processes to reduce the times and costs associated with robot-assisted laparoscopic radical prostatectomy. J Endourol. 2011 Jun;25(6):955-60. doi: 10.1089/end.2010.0534. Epub 2011 Apr 2. PMID 21457071
- [Background] de'Angelis N, Petrucciani N, Giannandrea G, Brunetti F. The protocol of low-impact laparoscopic cholecystectomy: the combination of mini-laparoscopy and low-pressure pneumoperitoneum. Updates Surg. 2018 Dec;70(4):553-556. doi: 10.1007/s13304-018-0591-8. Epub 2018 Aug 29. PMID 30159821